CLINICAL TRIAL: NCT04549272
Title: Assessment of Early Vascular Damage With Advanced Neuroimaging in Patient With Patent Foramen Ovale
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Giuseppe Lembo, Full Professor, MD, PhD, Neuromed IRCCS
Other Study IDs: LMB08
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Patent Foramen Ovale
Keywords: Magnetic Resonance Imaging; Vascular Cognitive Impairment
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Patent Foramen Ovale
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions - observational study

SUMMARY:
Patent foramen ovale arises from the incomplete postnatal fusion of the septum primum and secundum and can cause paradoxical embolism in adults. In case of cerebral ischemic stroke, the correlation with the patent foramen ovale is based on probabilistic approach. For this reason, continuous research is indispensable, especially according to new approaches, to offer tools capable of guiding in case of adverse event with greater certainty and even better to prevent it. Thus, this study aims to: 1) evaluate the microstructural brain damage through advanced MRI analysis in patients with patent foramen ovale; 2) evaluate how much the degree of the shunt can affect brain damage. In order to do this, this study aims to evaluate advanced brain imaging in a cohort of patients with patent foramen ovale to identify the development of early vascular damage.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 and ≤ 65 years
* patients with patent foramen ovale
* written informed consent

Exclusion Criteria:

* previous IMA, stroke or TIA
* arrhythmia or severe cardiac disease
* hypertension, diabetes or renal disease
* psychiatric disease
* neurological or neurodegenerative disease
* dementia
* assumption of drugs known to interfere with cognitive function
* inability to be subjected MRI analysis
* participation to other clinical trial, ongoing or terminated less than one month before enrolment in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from patients attending the Department of AngioCardioNeurology of the IRCCS Neuromed, accordingly to the following inclusion/exclusion criteria. Approximately 100 subjects of both genders will be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of percentage change in diffusion parameters of the white matter | At Enrollment
  Fiber tracking by DTI MRI

SECONDARY OUTCOMES:
Quantification of the degree of shunt of the patent foramen ovale | At Enrollment
  Echography
Detection of cognitive decline by decrease of MoCA score | At Enrollment
  Cognitive tests
Detection of a non-invasive retinal screening | At Enrollment
  Digital ophthalmoscope

IPD SHARING:
Plan to Share IPD: No